CLINICAL TRIAL: NCT03194178
Title: Impact of Phonatory and Facial Morphology Disorders, on the Quality of Life of Adolescents With Pierre Robin Sequence
Acronym: ADOROBIN
Status: Completed | Type: Observational
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMIS2016-01
Record Dates: First submitted 2017-06-09; First posted 2017-06-21 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Pierre Robin Syndrome
MeSH Terms: conditions — Pierre Robin Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pierre Robin sequence patients: Patients presenting a Pierre Robin sequence, and who have been cared in their early childhood by either the Necker or Trousseau hospitals teams, and who are between 12 and 18 years old at the beginning of the study.
  Interventions: Other: Pierre Robin sequence patients

INTERVENTIONS:
Other: Pierre Robin sequence patients — 4 questionnaires will be completed by the patient :
  * "Kidscreen 52" (generic quality of life questionnaire)
  * "Voice Handicap Index" : VHI-9i (specific quality of life questionnaire)
  * "Child Oral Health Impact Profile" : COHIP (specific quality of life questionnaire)
  * "MDI-C" (composite depression scale for minors)

SUMMARY:
The study team has made the hypothesis that the intensity of the phonatory disorders (rhinolalia), and of the maxillo-mandibular growth anomalies (facial morphology), may have negative effects on the quality of life of adolescents with Pierre Robin sequence.

The investigators also want to assess the impact of 2 different surgical protocols of closure of the cleft palate (1 or 2 step(s)), on the current phonatory and morphology aspects. These 2 protocols were performed, by 2 parisian clinical teams, that have now been merged at Necker hospital.

DETAILED DESCRIPTION:
In this protocol, the investigator will include patients who were treated, via maxillo-facial surgery, in their early childhood for a Pierre Robin sequence.

In the frame of a follow-up visit, if they accept to participate in the study, they will fulfill with 2 psychologists, 3 quality of life questionnaires, and 1 depression assessment questionnaire.

This will aim at evaluate their quality of life and their social integration, at the time of adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Having a Pierre Robin sequence, either isolated, either integrated to a collagenopathy, or associated to any other malformation, but without any mental retardation
* Being schooled in normal environment, with a maximum of 2 years of academic delay
* Having being treated, in the early childhood, for a maxillo-facial surgery, either in Paris-Necker or Paris-Trousseau hospitals (1 or 2 step(s) protocols)

Exclusion Criteria:

* Having any other form of Pierre Robin sequence (syndromic or associated to a mental retardation)
* Having more than 2 years of academic delay, or being schooled in a specialized environment
* Having an organic severe intercurrent disease, that could have an impact on the quality of life of the patients.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patient included will be patients affected with Pierre Robin sequence, and coming at the study reference center in the frame of a routine follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Correlation between generic and specific quality of life of the patients, scored via the questionnaires, and the severity of the troubles (facial and phonatory), assessed by the physicians | 3 years
  The data obtained via the 4 quality of life questionnaires will be assessed on regards of the severity of the facial dysmorphy and phonatory disorders.
  The investigators will aggregate these results, and will be able to check if there is a clear correlation between them. They will be able to say if it can be concluded that the physical troubles due to the Pierre Robin sequence affect the quality of life of the patients.

SECONDARY OUTCOMES:
Comparison of the generic quality of life of patients with Pierre Robin sequence, scored via the "Kidscreen 52" questionnaire, with the data of the general population | 3 years
  The investigator will assess the generic quality of life of the study patients, scored via the "Kidscreen 52" questionnaire, on regards of general population (data of the literature)
Comparison of the results of the 2 surgical protocols on the maxillo-mandibular growth | 3 years
  The investigator will compare the long-term maxillo-mandibular growth of the "Pierre Robin" patients, compared to the general population, and compared between the 2 surgical protocols used.
Comparison of the results of the 2 surgical protocols on the phonatory aftereffects | 3 years
  The investigator will compare the phonatory aftereffects of the "Pierre Robin" patients, compared to the general population, and compared between the 2 surgical protocols used.
Need of secondary surgery | 3 years
  The investigators will assess the need to realize a secondary surgery, according the initial surgery protocol used.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Abadie, Pr, Principal Investigator — Necker - Enfants Malades Hospital
Locations (1):
- Necker - Enfants Malades hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No